CLINICAL TRIAL: NCT04730310
Title: Association of Anesthesia Technique With Graft Patency Rates After Open Lower Limb Revascularization: a Retrospective Population Cohort Study
Brief Title: Anesthesia Technique and Lower Limb Revascularization Patency
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Prabhakar, Clinical Assistant Professor, Deparment of Anesthesiology, Pharmacology and Therapeutics, University of British Columbia
Other Study IDs: H20-03437
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Regional Anesthesia, Vascular Grafting, Vascular Patency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regional Anesthesia (RA): RA
  * Includes spinal, epidural, peripheral nerve block, excludes local infiltration (unlikely that any major open revascularization can be done under local)
  * Defined as: NSQIP Principal (ANESTHES) or additional (ANESTHES_OTHER) anesthesia technique = regional, spinal, epidural, or MAC (in NSQIP RA/Spinal/Local + MAC are coded as MAC; while this includes local + MAC, it would be unlikely that local anesthesia would be sufficient for open revascularization)
  Interventions: Procedure: NSQIP Lower Extremity Open (LEO) procedure-targeted dataset (i.e. undergoing Lower extremity open revascularization) from 2014-2019
- General Anesthesia (GA): GA
  * Defined as: NSQIP Principal or additional anesthesia technique = general
  * Since GA is selected as the principal anesthetic technique by default when multiple techniques are present, GA + RA could potentially have been coded as GA if the optional variable of additional anesthesia technique is not filled in, leading to differential misclassification of patients with GA + RA (most likely epidural and peripheral nerve block) in the GA group.
  Interventions: Procedure: NSQIP Lower Extremity Open (LEO) procedure-targeted dataset (i.e. undergoing Lower extremity open revascularization) from 2014-2019

INTERVENTIONS:
Procedure: NSQIP Lower Extremity Open (LEO) procedure-targeted dataset (i.e. undergoing Lower extremity open revascularization) from 2014-2019 — Infrainguinal, open lower extremity revascularization procedures

SUMMARY:
The role of regional anesthesia in lower extremity revascularization procedures on reducing graft failure and need for reoperation remains unclear. In this study, we will analyze data from the multicenter National Surgical Quality Improvement Program (ACS NSQIP®) to assess the association between regional anesthesia (RA) and graft outcomes, as compared to general anesthesia (GA). Our primary objective is to determine for patients undergoing elective open lower limb revascularization, whether RA (spinal, epidural, and peripheral nerve block), compared to GA or general anesthesia with regional anesthesia (GA+RA), is associated with higher rates of patent graft within 30 days postoperatively (primary outcome).

DETAILED DESCRIPTION:
Lower limb (infrainguinal) revascularization surgeries are performed for patients with blood flow occlusion, with the goals of improving pain and function. Graft patency is associated with higher quality of life scores. However, open lower limb revascularization is associated with a significant risk of graft failure. Multiple anesthesia options exist for elective open lower limb revascularization, including general and regional (spinal, epidural, peripheral nerve block). The literature has shown mixed results regarding the superiority of regional anesthesia over general anesthesia for morbidity and mortality. In this study, we will analyze data from the multicenter National Surgical Quality Improvement Program (ACS NSQIP®) to assess the association between regional anesthesia (RA) and graft outcomes, as compared to general anesthesia (GA).Our primary objective is to determine for patients undergoing elective open lower limb revascularization, whether RA (spinal, epidural, and peripheral nerve block), compared to GA or general anesthesia with regional anesthesia (GA+RA), is associated with higher rates of patent graft within 30 days postoperatively (primary outcome). Our secondary outcomes are major reintervention, amputation, bleeding requiring transfusion or secondary procedure, venous thromboembolism (VTE), myocardial infarction (MI) or stroke, pneumonia, discharge destination, postoperative length of stay, readmission rate, and death, all within 30 days postoperatively. There will be two composite outcomes: thromboembolism, and morbidity and mortality. We hypothesize that the use of RA is associated with increased graft patency after elective lower limb revascularization compared to GA. Compared to GA, RA is associated with decreased rates of major reintervention, amputation, death (30 days), bleeding requiring transfusion or secondary procedure, VTE, MI or stroke, pneumonia, mortality, composite thromboembolism, and composite morbidity and mortality.; Compared to GA, RA is associated with increased rates of discharge destination being home.

ELIGIBILITY:
Inclusion Criteria:

* All elective cases within the NSQIP Lower Extremity Open (LEO) procedure-targeted dataset (i.e. undergoing Lower extremity open revascularization) from 2014-2019 will be included.
* Hybrid procedures (where patients had both open and endovascular repair) are included, as long as there is an open component.

Exclusion Criteria:

* Patients will be excluded if they underwent urgent or emergency surgery (identified using NSQIP variable EMERGNCY=1 OR ELECTSURG=0)
* local was the only anesthetic technique listed in principal and additional anesthesia technique.
* missing data on exposure, procedure name, or status of elective surgery. This includes having "other" or "unknown" for BOTH principal and additional anesthesia technique
* Patients with INR >= 1.5 on day of surgery

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All elective cases within the NSQIP Lower Extremity Open (LEO) procedure-targeted dataset (i.e. undergoing Lower extremity open revascularization) from 2014-2019 will be included. The estimated sample size is 15,000 based on the NSQIP Participant Use Files.
  Elective procedures will be identified using the NSQIP variable ELECTSURG=1. Urgent and emergency procedures are not included, as patients may not being offered RA due to insufficient time and/or unable to withhold anticoagulants/antiplatelets due to acute limb ischemia. Note that age 18 years and older is already part of the NSQIP inclusion criteria. Hybrid procedures (where patients had both open and endovascular repair) are included, as long as there is an open component.
Sampling Method: Probability Sample
Enrollment: 8893 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Graft Patency | 30 days
  * Derived using NSQIP variables "Most Severe Procedural Outcome" LEO_MOSTSEVOUTCOME and "Untreated Loss of Patency" (i.e. not patent and no procedure done) LEO_ULP
  * Yes if LEO_MOSTSEVOUTCOME is any of
  * Clinically Patent Graft
  * Patent graft, no stenosis
  * Patent graft with stenosis
  * No if LEO_MOSTSEVOUTCOME is any of
  * Death
  * Image-proven graft thrombosis or clinically evident thrombosis with no planned intervention
  * Major Amputation
  * New bypass in the treated arterial segment
  * Not documented
  * Other
  * Revised graft with stenosis
  * Revised graft, no current stenosis
  * No if LEO_ULP = "yes"

SECONDARY OUTCOMES:
Major reintervention | 30 days
  1. Major reintervention, using NSQIP variable "Major Reintervention on the Bypass" defined as ""Yes" if the patient underwent a subsequent procedure (new or revision lower extremity bypass operation, jump/interposition graft revision, bypass graft thrombectomy/thrombolysis) within 30 days of the original primary operation."
Amputation | 30 days
  2. Amputation, using NSQIP variable "Major Amputation (Transtibial or Proximal)", defined as ""Yes" if the patient underwent transtibial or more proximal amputation on the ipsilateral leg within 30 days of the original primary operation."
Bleeding requiring transfusion | 30 days
Venous thromboembolism | 30 days
MI or stroke | 30 days
Pneumonia | 30 days
length of postoperative hospital stay | 30 days
Discharge destination | 30 days
  dichotomize as home vs. not home
Readmission rate | 30 days
death | 30 days or in-hospital admission
Composite thromboembolism | 30 days
  combination of venothromboembolism, MI, stroke
Composite Morbidity and Mortality | 30 days
  combination of bleeding requiring transfusion, venothromboembolism, MI, stroke, pneumonia, death

OTHER OUTCOMES:
Confounders | day of surgery
  age, bleeding diathesis, severe COPD, total operating, time, renal failure, functional status, cardiac valvular disease, diabetes
Confounders | day of surgery
  INR, PTT

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
NSQIP data would be free to other researchers from central site.

REFERENCES:
- [Background] Barbosa FT, Juca MJ, Castro AA, Cavalcante JC. Neuraxial anaesthesia for lower-limb revascularization. Cochrane Database Syst Rev. 2013 Jul 29;2013(7):CD007083. doi: 10.1002/14651858.CD007083.pub3. PMID 23897485
- [Background] Nguyen LL, Moneta GL, Conte MS, Bandyk DF, Clowes AW, Seely BL; PREVENT III Investigators. Prospective multicenter study of quality of life before and after lower extremity vein bypass in 1404 patients with critical limb ischemia. J Vasc Surg. 2006 Nov;44(5):977-83; discussion 983-4. doi: 10.1016/j.jvs.2006.07.015. PMID 17098529
- [Background] Grip O, Wanhainen A, Michaelsson K, Lindhagen L, Bjorck M. Open or endovascular revascularization in the treatment of acute lower limb ischaemia. Br J Surg. 2018 Nov;105(12):1598-1606. doi: 10.1002/bjs.10954. Epub 2018 Jul 25. PMID 30043994
- [Background] Ghanami RJ, Hurie J, Andrews JS, Harrington RN, Corriere MA, Goodney PP, Hansen KJ, Edwards MS. Anesthesia-based evaluation of outcomes of lower-extremity vascular bypass procedures. Ann Vasc Surg. 2013 Feb;27(2):199-207. doi: 10.1016/j.avsg.2012.04.006. Epub 2012 Sep 1. PMID 22944010
- [Background] Sgroi MD, McFarland G, Mell MW. Utilization of regional versus general anesthesia and its impact on lower extremity bypass outcomes. J Vasc Surg. 2019 Jun;69(6):1874-1879. doi: 10.1016/j.jvs.2018.08.190. Epub 2019 Feb 18. PMID 30792062
- [Background] Fereydooni A, O'Meara T, Popescu WM, Dardik A, Ochoa Chaar CI. Utilization and Outcomes of Local Anesthesia and Peripheral Nerve Block for Hybrid Lower Extremity Revascularization. J Endovasc Ther. 2020 Feb;27(1):94-101. doi: 10.1177/1526602819887382. Epub 2019 Nov 20. PMID 31746264
- [Background] Roberts DJ, Nagpal SK, Kubelik D, Brandys T, Stelfox HT, Lalu MM, Forster AJ, McCartney CJ, McIsaac DI. Association between neuraxial anaesthesia or general anaesthesia for lower limb revascularisation surgery in adults and clinical outcomes: population based comparative effectiveness study. BMJ. 2020 Nov 25;371:m4104. doi: 10.1136/bmj.m4104. PMID 33239330
- [Background] Christopherson R, Beattie C, Frank SM, Norris EJ, Meinert CL, Gottlieb SO, Yates H, Rock P, Parker SD, Perler BA, et al. Perioperative morbidity in patients randomized to epidural or general anesthesia for lower extremity vascular surgery. Perioperative Ischemia Randomized Anesthesia Trial Study Group. Anesthesiology. 1993 Sep;79(3):422-34. doi: 10.1097/00000542-199309000-00004. PMID 8363066
- [Background] Wiis JT, Jensen-Gadegaard P, Altintas U, Seidelin C, Martusevicius R, Mantoni T. One-week postoperative patency of lower extremity in situ bypass graft comparing epidural and general anesthesia: retrospective study of 822 patients. Ann Vasc Surg. 2014 Feb;28(2):295-300. doi: 10.1016/j.avsg.2013.01.027. Epub 2013 Sep 29. PMID 24084268
- [Background] Jorgensen MS, Farres H, James BLW, Li Z, Almerey T, Sheikh-Ali R, Clendenen S, Robards C, Erben Y, Oldenburg WA, Hakaim AG. The Role of Regional versus General Anesthesia on Arteriovenous Fistula and Graft Outcomes: A Single-Institution Experience and Literature Review. Ann Vasc Surg. 2020 Jan;62:287-294. doi: 10.1016/j.avsg.2019.05.016. Epub 2019 Aug 2. PMID 31382001
- [Background] Gao C, Weng C, He C, Xu J, Yu L. Comparison of regional and local anesthesia for arteriovenous fistula creation in end-stage renal disease: a systematic review and meta-analysis. BMC Anesthesiol. 2020 Aug 31;20(1):219. doi: 10.1186/s12871-020-01136-1. PMID 32867692
- [Background] Goodney PP, Nolan BW, Schanzer A, Eldrup-Jorgensen J, Bertges DJ, Stanley AC, Stone DH, Walsh DB, Powell RJ, Likosky DS, Cronenwett JL; Vascular Study Group of Northern New England. Factors associated with amputation or graft occlusion one year after lower extremity bypass in northern New England. Ann Vasc Surg. 2010 Jan;24(1):57-68. doi: 10.1016/j.avsg.2009.06.015. Epub 2009 Sep 11. PMID 19748222
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839